CLINICAL TRIAL: NCT05320510
Title: Effect of Selenium Supplementation on Glycemic Control in Patients With Type 2 Diabetes or Prediabetes: a Double Blinded, Randomized Controlled Trail
Brief Title: Effect of Selenium Supplementation on Glycemic Control in Patients With Type 2 Diabetes or Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LK20220322
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes; PreDiabetes
Keywords: selenium; Type 2 Diabetes; prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Se-yeast (Experimental): Selenium-enriched yeast tablet (Se, 50 μg/d)
  Interventions: Dietary Supplement: Se-yeast
- Placebo (Placebo Comparator): placebo-yeast tablet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Se-yeast — The participants will be asked to take Se-yeast tablet. The intervention period is about 3 months. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Se-yeast
Dietary Supplement: Placebo — The participants will be asked to take placebo-yeast tablet. The intervention period is about 3 months. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Placebo

SUMMARY:
Although it has been suggested that selenium (Se) increases the risk of T2DM, most evidence comes from observational studies that cannot prove causality. A systematic review assessed randomized clinical trials and found that the risk of T2DM was not greater in those randomized to Se supplementation than in those randomized to placebo. Se is a toxic element in animals and humans, and overexposure to Se has also been linked to detrimental health effects in humans. Previous studies were mostly conducted in Se-sufficient areas. Moreover, the effectiveness of low-dose Se supplementation on participants with elevated glycemic status was unknown. This cross-over, double blinded, randomized controlled trail aimed to investigate the effectiveness of Se supplementation for glucose control among participants with diabetes or prediabetes. Moreover, we also aimed to examine whether selenoprotein P genotypes, Se-related gut microbiota and their related metabolite modified the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. FPG ≥ 5.6 mmol/L;
2. HbA1c ≥ 5.7%;
3. OGTT 2h or postprandial blood glucose ≥ 7.8 mmol/L.
4. T2D patients with stable anti-diabetic medication and blood glucose controlled well for 4 weeks prior.

Exclusion Criteria:

1. Under 30 years old or above 70 years old;
2. Pregnancy;
3. Major surgery in the previous 6 months or planned to occur during the trail;
4. Insulin injection for diabetes;
5. Suffering from severe obesity (BMI > 40 kg/m2), immunodeficiency syndrome, thyroid disease, coronary heart disease, stroke, malignant neoplasm, kidney or liver disease, or other serious diseases, such as mental illness;
6. Reduced kidney function (GFR < 60 mL/min/1.73m2, creatinine > 1.2 times the normal upper limit [male, > 133.2 μmol/L; female > 100 μmol/L]);
7. Systolic or diastolic blood pressure greater than 160 or 100 mmHg;
8. Taking dietary supplements (e.g., selenium, vitamin, fish oil, etc.) for nearly one month before the intervention;
9. Taking antibiotics or probiotics within 12 weeks of screening.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c concentration | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of glycated hemoglobin concentration

SECONDARY OUTCOMES:
Change of FPG concentration | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of fasting plasma glucose concentration
Change of FPI concentration | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of fasting plasma insulin concentration
Change of HOMA-IR | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of homeostasis model of assessment-insulin resistance
Change of TG concentration | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of serum triglyceride concentration
Change of TC concentration | 0 week, 4th week, 8th week, and 12th week in the intervention period
  Change of total cholesterol concentration

IPD SHARING:
Plan to Share IPD: No